CLINICAL TRIAL: NCT05903404
Title: The PCOS Indirect and Intangible Economic Burden Study. A Sub-study of the PCOS Challenge Study: For the Collection of Information to Advance Research and Improve Care for PCOS Patients
Brief Title: PCOS Indirect and Intangible Economic Burden
Acronym: PCOSCHALLENGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PCOS Challenge: The National Polycystic Ovary Syndrome Association (Other)
Responsible Party: Sponsor
Other Study IDs: PCOSC002: PCOS Economic Burden
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: pcos; polycystic ovary syndrome; polycystic ovarian syndrome; stein leventhal syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Target Population: The target population includes individuals diagnosed with PCOS by a healthcare provider, self-diagnosed with PCOS, or who are exhibiting PCOS Symptoms and willing to sign the consent.
- Control Population: The control population includes people born biologically female who have not been diagnosed with PCOS and who also do not have symptoms of PCOS.

SUMMARY:
The primary purpose of the PCOS Indirect and Intangible Economic Buren study is to estimate the economic costs of having PCOS in terms of quality of life and work productivity. The population will include individuals with a clinical diagnosis of PCOS, individuals self-diagnosed with PCOS, individuals with symptoms of PCOS (e.g., hirsutism, irregular menstrual cycles), and demographic-matched controls without PCOS. This study is a sub-study of The PCOS Challenge Study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PCOS by a health professional, self-diagnosed with PCOS or individuals with PCOS symptoms
* Willing to sign the consent form
* Able to understand the registry surveys or what is being asked

Exclusion Criteria:

* Unable to understand the surveys or what is being asked
* Unwilling to sign the consent form

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Born biologically female
Study Population: The population for the PCOS Indirect and Intangible Economic Burden will include individuals with a clinical diagnosis of PCOS, individuals self-diagnosed with PCOS, individuals with symptoms of PCOS (e.g., hirsutism, irregular menstrual cycles), and demographic-matched controls without PCOS.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Information | One Year
  Such as responses to survey questions

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Ottey, MHA, MT (ASCP), Principal Investigator — PCOS Challenge: The National Polycystic Ovary Syndrome Association; Ricardo Azziz, MD, MPH, MBA, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- PCOS Challenge: The National Polycystic Ovary Syndrome Association, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in PCOS. Data or samples shared will be coded, with no PHI included.
Supporting Information: Study Protocol